CLINICAL TRIAL: NCT03829384
Title: A Phase 1, Randomized, Placebo-Controlled, Dose Ranging Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of mRNA-1944, Encoding for an Anti-Chikungunya Virus Monoclonal Antibody, in Healthy Adults
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of mRNA-1944 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1944-P101
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Prevention of Chikungunya Virus Infection
Keywords: Chikungunya fever; Alphavirus infections; Togavirus; Viral diseases
MeSH Terms: conditions — Chikungunya Fever; Alphavirus Infections; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mRNA-1944 (Experimental): Escalating dose levels
  Interventions: Biological: mRNA-1944
- Placebo (Placebo Comparator): Saline
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: mRNA-1944 — mRNA encoding Chikungunya antibody
  Arms: mRNA-1944
Other: Placebo — Saline
  Arms: Placebo

SUMMARY:
This is a Phase 1, FIH, single-center, randomized, placebo controlled, dose escalation study to evaluate the safety, tolerability, PK, and PD of mRNA-1944 in healthy adult subjects. Cohorts of mRNA-1944 are planned to be investigated in a sequential dose escalation manner.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 and ≤ 50 years of age
* Weight of 50 to 100 kg, inclusive
* In good general health as determined by medical history, clinical laboratory assessments, ECG results, vital sign measurements, and physical examination findings at screening
* Has access to consistent and reliable means of contact and agrees to stay in contact with the study site for the duration of the study

Exclusion Criteria:

* Any acute or chronic clinically significant disease, as determined by physical examination or laboratory screening tests
* Elevated liver function tests or safety laboratory test results
* Positive screening test for the presence of anti-CHIKV IgG
* Administration of another investigational study involving any investigational product within 60 days or 5 half-lives, whichever is longer
* Has received any live attenuated or inactive vaccines within 4 weeks prior to check-in, or plans to receive any vaccine during the study
* Known or suspected immune-mediated disease or immunosuppressive condition (including lymphoproliferative disorders)
* Any neurologic disorder
* History of idiopathic urticaria
* Any bleeding disorder that is considered a contraindication to study drug infusion or blood collection
* Receipt of immunoglobulins, a monoclonal antibody or any blood products within the preceding 6 months
* Any acute illness at the time of enrollment
* A positive test result for drugs of abuse
* A positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus type 1 or 2 antibodies
* A history of active cancer (malignancy) in the last 3 years
* Donation of ≥ 450 mL blood or blood products within 30 days of study drug infusion

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs), serious adverse events (SAEs), adverse events of special interest (AESI) and laboratory abnormalities | Through 13 months of study participation

SECONDARY OUTCOMES:
Area under the concentration versus time curve (AUC) | Baseline through 28 days post dose
Maximum observed serum concentration (Cmax) after administration of mRNA-1944 | Baseline through 28 days post dose
Time of Cmax (tmax) | Baseline through 28 days post dose
Terminal elimination half-life (t1/2) | Baseline through 28 days post dose
Maximum observed effect (Emax) for chikungunya virus IgG | Baseline through 13 months
Time to maximum observed effect for (TEmax) for chikungunya virus IgG | Baseline through 13 months
Area under the effect curve (AUEC) for chikungunya virus IgG | Baseline through 13 months

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Phase 1 Clinical Research Unit, Austin, Texas, United States

REFERENCES:
- [Derived] Deng YQ, Zhang NN, Zhang YF, Zhong X, Xu S, Qiu HY, Wang TC, Zhao H, Zhou C, Zu SL, Chen Q, Cao TS, Ye Q, Chi H, Duan XH, Lin DD, Zhang XJ, Xie LZ, Gao YW, Ying B, Qin CF. Lipid nanoparticle-encapsulated mRNA antibody provides long-term protection against SARS-CoV-2 in mice and hamsters. Cell Res. 2022 Apr;32(4):375-382. doi: 10.1038/s41422-022-00630-0. Epub 2022 Feb 24. PMID 35210606
- [Derived] August A, Attarwala HZ, Himansu S, Kalidindi S, Lu S, Pajon R, Han S, Lecerf JM, Tomassini JE, Hard M, Ptaszek LM, Crowe JE, Zaks T. A phase 1 trial of lipid-encapsulated mRNA encoding a monoclonal antibody with neutralizing activity against Chikungunya virus. Nat Med. 2021 Dec;27(12):2224-2233. doi: 10.1038/s41591-021-01573-6. Epub 2021 Dec 9. PMID 34887572